CLINICAL TRIAL: NCT04173715
Title: Validation of Cut-points to Estimate Sedentary Time and Physical Activity Intensities in Older Adults
Brief Title: Movement and Behaviours Measurement Study
Acronym: MOBEMENTS
Status: Recruiting | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Ignacio Ara, Associate Professor, University of Castilla-La Mancha
Other Study IDs: CEIC-CHT-568
Record Dates: First submitted 2019-10-31; First posted 2019-11-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Aging; Physical Function; Frailty Syndrome; Physical Disability; Lifestyle, Sedentary
Keywords: Cut-Points; Accelerometry; Physical Activity Quantification; Physical Function; Frailty Syndrome; Energy Expenditure; Aging
MeSH Terms: conditions — Frailty; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- General Group: All those who are over 65 years old and capable of walking by themselves.
  Interventions: Behavioral: Older Adults Group.
- Low Physical Function Status Group.: All those who present a low physical function status will be included in this group.
  Interventions: Behavioral: Low Physical Function Status Group; Behavioral: Medium Physical Function Status Group
- Medium Physical Function Status Group.: All those who present a medium physical function status will be included in this group.
  Interventions: Behavioral: Low Physical Function Status Group; Behavioral: Medium Physical Function Status Group; Behavioral: High Physical Function Status Group
- High Physical Function Status Group.: All those who present a high physical function status will be included in this group.
  Interventions: Behavioral: High Physical Function Status Group

INTERVENTIONS:
Behavioral: Older Adults Group. — Physical activity and energy expenditure quantification
  Groups: General Group
Behavioral: Low Physical Function Status Group — Physical activity and energy expenditure quantification
  Groups: Low Physical Function Status Group.; Medium Physical Function Status Group.
Behavioral: Medium Physical Function Status Group — Physical activity and energy expenditure quantification
  Groups: Low Physical Function Status Group.; Medium Physical Function Status Group.
Behavioral: High Physical Function Status Group — Physical activity and energy expenditure quantification
  Groups: High Physical Function Status Group.; Medium Physical Function Status Group.

SUMMARY:
There are few studies that already have validated specific raw accelerometer cut-points for people over 65 years old.

The purpose of the present study is to validate raw accelerometer cut points for general people over 65 years old and specific raw accelerometer cut points based on the functional status of older adults over 65 years old.

The study will be carried out with an observational approach. Participants will be divided into 4 groups. First of them will be made grouping all subjects and the rest divided according to their functional status. They will perform different-intensity physical activities while wearing accelerometers attached to their body and wearing a portable gas analyser too. Their intensity will be assessed based on their own Rest Metabolic Rate (RMR). Energy expenditure and accelerations will be matched and, based on that, sedentary behaviour, light physical activity and moderate-to-vigorous physical activity cut-points will be derived.

DETAILED DESCRIPTION:
Knowledge on health implications of sedentary time and physical activity has been substantially improved in the last decades with accelerometer-based estimations. The popularity of these devices is partially explained by the capacity of objectively recording physical behaviors (e.g., sleep, sedentary time, physical activity…) during the whole day. The so-called "cut-point" approach is behind most of the research on physical activity with accelerometers. Cut-points provide metrics that are easy to understand, to translate to the public and to replicate by researchers in different settings. Usually, the minimum requirement is to use cut-points adapted to the age-group of the population of interest.

Under this paradigm, cut-points have been developed in all age-groups and with a variate set to data collection and processing protocols. However, some scenarios lack of available cut-points to implement, being older adults (> 65 years) the population with less alternatives of cut-points to use. In this sense, studies with older adults choose cut-points developed in younger adults to classify physical activity intensities. Biomechanical and physiological differences between adults and older adults advise against using this strategy. Therefore, relative energy expenditure and functional status should be considered for future cut-points design. Moreover, must be also awarded that hardly any previous cut-points validation protocols have been performed in a free-living setting. For this reason, more studies following these designs seems necessary to improve cut-points population's validity. Missing all mentioned factors could lead to physical activity and sedentary behavior patterns misclassification in this population.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* Non-institutionalized
* Physical function assessment (SPPB>3)

Exclusion Criteria:

* Have started an exercise program.
* Mini-Mental Score < 18.
* Presenting any physical activity contraindication.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: People over 65 years old will be enrolled in the study. They will be recruited from the Frailty Consultation in the Virgen del Valle Hospital from Toledo (Spain).
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-10-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Rest Metabolic Rate | Through study completion, an average of 1 year
  (ml/kg-1/min-1)
Energy expenditure during physical activity performance | Through study completion, an average of 1 year
  (ml/kg-1/min-1)
Accelerometry | Through study completion, an average of 1 year
  Gravitational Units
Physical function | Through study completion, an average of 1 year
  Short Physical Performance Battery
Frailty Status | Through study completion, an average of 1 year
  Fried Frailty Index (0 criteria: Robust; 1-2 criteria: Pre-frail; >2 criteria: Frail) and Frailty Trait Scale (from 0 (best score) to 100 (worst score))
Physical Activity and Sedentary Behaviour Patterns. | Through study completion, an average of 1 year
  Accelerometers

SECONDARY OUTCOMES:
Heart Rate | Through study completion, an average of 1 year
  (bpm)
Body composition | Through study completion, an average of 1 year
  Dual energy X-ray Absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Ara Royo, Principal Investigator — Univeristy of Castilla-La Mancha
Locations (1):
- Universidad de Castilla-La Mancha, Laboratorio de Actividad Física y Función Muscular, Toledo, Spain